CLINICAL TRIAL: NCT01113619
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effectiveness, Safety and Tolerability of RP-G28 in Subjects With Symptoms Associated With Lactose Intolerance
Brief Title: Effectiveness, Safety and Tolerability Study of RP-G28 for Symptoms Associated With Lactose Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ritter Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G28-001
Record Dates: First submitted 2010-04-23; First posted 2010-04-30 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Lactose Intolerance
Keywords: lactose maldigestion; dairy intolerance; intolerance to milk; intolerance to dairy; milk intolerance; GI disorder; lactose metabolism; GI symptoms after dairy ingestion
MeSH Terms: conditions — Lactose Intolerance | interventions — RP-G28

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RP-G28 (Experimental): Study Drug RP-G28
  Interventions: Drug: RP-G28 or placebo
- Placebo (Placebo Comparator): Study Drug Placebo
  Interventions: Drug: RP-G28 or placebo

INTERVENTIONS:
Drug: RP-G28 or placebo — Qualified subjects randomized to daily dosing with RP-G28 or placebo
Drug: RP-G28 or placebo — Daily dosing

SUMMARY:
This is a Phase 2 study designed to assess the ability of RP-G28 to improve lactose digestion and tolerance.

DETAILED DESCRIPTION:
Lactose intolerance is a common gastrointestinal (GI) disorder that develops in lactose maldigesters when consuming too much lactose or when lactose is added to a previously low-lactose diet. Lactose intolerance is characterized by one or more of the cardinal symptoms that follow the ingestion of lactose-containing foods. These symptoms include; abdominal pain/cramps, bloating, flatulence [gas] and diarrhea. As such, most lactose intolerant individuals avoid the ingestion of milk and dairy products, while others substitute non-lactose containing products in their diet.

Based on the health implications from insufficient calcium intake over a lifetime, including increased risk of osteoporosis and hypertension, there is need in the medical community for a tolerable and convenient treatment that allows for all levels of milk and dairy product consumption in people suffering from mild to severe lactose intolerance. This study will evaluate a treatment that provides a simplified dosing regimen as well as the potential for extended relief from symptoms following a limited therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects. Female subjects must be non-pregnant and non-lactating.
* 18 to 64 years of age inclusive at Screening
* Current or recent history of intolerance to milk and other dairy products
* Acceptable Baseline Lactose Intolerance Symptom Scores
* Acceptable Result on Baseline Hydrogen Breath Test
* Subjects must agree to refrain from all other treatments and products used for lactose intolerance during the study

Exclusion Criteria:

* Disorders known to be associated with abnormal GI motility
* History of surgery that alters the normal function of the gastrointestinal tract
* Past or present; organ transplant, chronic pancreatitis, pancreatic insufficiency, symptomatic biliary disease, Celiac disease, inflammatory bowel disease (IBD), ulcerative colitis, Crohn's disease, irritable bowel syndrome (IBS)
* Active gastric or duodenal ulcers or history of severe ulcers
* Diabetes mellitus (type 1 or type 2)
* Congestive Heart Failure
* History of Human Immunodeficiency Virus (HIV), Hepatitis B or C
* Use of concurrent therapy(ies) for symptoms of lactose intolerance
* Uncontrolled BP defined as sitting systolic blood pressure (SBP) ≥160 mmHg or diastolic blood pressure (DBP) ≥95 mmHg at Visit 1
* History of ethanol abuse in the past 12 months
* History of drug abuse within 12 months
* History or presence of malignancy within the past 5 years (except basal cell or squamous cell carcinoma removed from a sun-exposed area)
* Use of any investigational drug or participation in any investigational study within 30 days prior to Screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
1) Change from Baseline in breath hydrogen production on Hydrogen Breath Test. 2) Change from Baseline in lactose intolerance symptom assessment during lactose challenge | Baseline, 36 days

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as Measure of Safety and Tolerability | 36 days
  Number of Subjects with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Covance, Inc. - Honolulu, Honolulu, Hawaii
  - Covance, Inc. - Dallas, Dallas, Texas

REFERENCES:
- [Derived] Savaiano DA, Ritter AJ, Klaenhammer TR, James GM, Longcore AT, Chandler JR, Walker WA, Foyt HL. Improving lactose digestion and symptoms of lactose intolerance with a novel galacto-oligosaccharide (RP-G28): a randomized, double-blind clinical trial. Nutr J. 2013 Dec 13;12:160. doi: 10.1186/1475-2891-12-160. PMID 24330605